CLINICAL TRIAL: NCT03473782
Title: Overactive Bladder (OAB) Voiding Diary and Urodynamics Correlation Study
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 15-00827
Record Dates: First submitted 2018-03-16; First posted 2018-03-22 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Voiding Diary
  Interventions: Other: Voiding Diary; Other: Urodynamics Correlation Study
- Urodynamics Correlation Study
  Interventions: Other: Voiding Diary; Other: Urodynamics Correlation Study

INTERVENTIONS:
Other: Voiding Diary — A log kept by each patient to record frequency and volume of urine output and fluid input.
Other: Urodynamics Correlation Study — Provides patho physiological data by assessing bladder sensation, bladder capacity, the presence of involuntary bladder contractions, bladder compliance and bladder outlet obstruction.

SUMMARY:
This is a prospective cohort study study with the primary aim of identifying the strongest correlating parameters between voiding diaries and UDS studies most predictive for each type of urologic condition. Investigators will focus on OAB related conditions, as these are symptoms

ELIGIBILITY:
Inclusion Criteria:

* completing a bladder diary
* undergoing VUDS

Exclusion Criteria:

* have a urinary tract infection
* neurogenic bladder
* history of pelvic irradiation
* prolapse alone without LUTS
* pregnant
* incarcerated
* hospital employee
* unable to give consent

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen regularly with Overactive Bladder (OAB)
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2015-10-12 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Measure of urgency incontinence using Voiding Diary | 60 Months
  patients will record urgency in diary

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Brucker, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States